CLINICAL TRIAL: NCT05867849
Title: Cannabidiol Adjunctive Therapy for Acute Bipolar Depression: A Randomized Double-Blind, Placebo Controlled Trial
Brief Title: Cannabidiol for Bipolar Depression (CBD-BD)
Acronym: CBD-BD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lakshmi N Yatham, Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H23-00105
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Disorder
Keywords: Cannabidiol; Bipolar Disorder; Bipolar Depression; Mood Disorder; CBD; Depression
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Cannabidiol 200 - 600 mg / day added to current treatment for 6 weeks.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Placebo added to current treatment for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Cannabinoid
  Other Names: CBD
  Arms: Cannabidiol
Other: Placebo — Inactive substance
  Arms: Placebo

SUMMARY:
Bipolar disorder (BD) is a lifelong condition characterized by recurrent episodes of depression and (hypo)mania. Periods of chronic and recurring depressive episodes are more common and can be severely disabling. Effective treatments exist; however, a significant portion of bipolar depressed patients do not respond to or have difficulty tolerating many of these interventions and thus look beyond established treatments to achieve symptom relief.

Cannabidiol (CBD), a chemical from the Cannabis sativa plant, has shown to have some beneficial effects on mood symptoms in a few small studies which assessed its effects in other mental and physical health conditions, but no large studies have been conducted to assess its safety and efficacy in bipolar depression. Additionally, several clinical studies have shown CBD to be safe and tolerable.

The primary objective of this study is to assess the effectiveness, safety and tolerability of cannabidiol in patients with bipolar depression (BD I or BD II) who have not responded to adequate trials with at least one first-line treatment for bipolar depression in comparison to those who will be treated with placebo. Placebo is an inactive substance that looks identical to the study medication but contains no therapeutic ingredient. This study is a randomized (like the flip of a coin), double-blind (you and the study team will not know which treatment arm you receive) study in which participants will receive either CBD or placebo added to their current treatment. Participants will have 5 clinical appointments and a phone appointment over a period of 10 weeks.

DETAILED DESCRIPTION:
This is a Phase 3, 6-week, double-blind, parallel group randomized controlled trial to assess the efficacy, safety and tolerability of adjunctive CBD vs placebo in patients with acute bipolar depression (BD I or BD II) who have not responded to adequate trials with at least one first-line treatment for bipolar I disorder (i.e. lithium, lamotrigine, lurasidone, or quetiapine either as monotherapy or adjunctive therapy), or at least one first or second-line treatment for bipolar II depression (i.e. quetiapine, lithium, lamotrigine, sertraline, or venlafaxine as monotherapy or adjunctive therapy, or bupropion adjunctive therapy). After the baseline visit, patients who meet the eligibility criteria will enter a 6-week double-blind treatment phase during which participants will be randomized to adjunctive CBD or identical placebo.

Participants will be assessed at the screening visit, baseline visit, weeks 2, 4, and 6, or endpoint visit. All participants will receive a follow-up telephone call 2 weeks after the 6-week study endpoint or early termination visit to assess well-being.

All participants will continue treatment with their mood stabilizer and/or atypical antipsychotic as prescribed by their treating physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 19 to 70 years (inclusive).
2. DSM-5 diagnosis of BD I or BD II, AND a current major depressive episode confirmed by MINI 7.0.2 .
3. All patients must be taking either a mood stabilizer (i.e. lithium or valproate; lamotrigine monotherapy as a mood stabilizer is acceptable for BD II patients only and not for BD I) OR an atypical antipsychotic OR a combination of these (two mood stabilizers or a mood stabilizer plus an atypical antipsychotic), at therapeutic doses. Medications and therapeutic doses are: lithium, serum level 0.6-1.2 mEq/L; divalproex/sodium valproate, serum level 350-700 uM/L(45-125 mcg/ml); risperidone 2-6 mg/day; olanzapine 5-30 mg/day; quetiapine IR or XR 300-900 mg/day; aripiprazole 10-30 mg/day; cariprazine 1.5-6 mg/day; and ziprasidone 80-160 mg/day. Combinations of these medications as outlined above, or the combination of any of them with lamotrigine 100-400 mg daily, or the combination of a mood stabilizer plus asenapine 5-20 mg/day are also permitted.
4. Have received a minimum of 6-weeks treatment at adequate doses for treatment of current depressive episode with at least one CANMAT recommended first-line treatment for bipolar I disorder (i.e. lithium, lamotrigine, lurasidone, or quetiapine either as monotherapy or adjunctive therapy), or at least one first or second-line treatment for bipolar II depression (i.e. quetiapine, lithium, lamotrigine, sertraline, or venlafaxine as monotherapy or adjunctive therapy, or bupropion adjunctive therapy).
5. A MADRS score of ≥ 20 and a YMRS score of ≤ 12 (these cut off scores are standard in bipolar depression RCTs).
6. Inpatient or outpatient status.
7. All participants are required to agree to practice highly effective methods of contraception (i.e. hormonal contraceptives, intrauterine device or system, vasectomy and tubal ligation, or double barrier methods of contraception) OR agree to completely abstain from heterosexual intercourse. Females who do not have childbearing potential are required to be postmenopausal for at least 1 year before the screening visit (confirmed by an FSH test) OR surgically sterile.
8. The capability of understanding, consenting to and complying with study requirements.
9. All concomitant medication must be at a stable dose for two weeks prior to the randomization visit.

Exclusion Criteria:

1. Current depressive episode greater than 12 months.
2. A history of rapid cycling, defined as ≥ 4 mood episodes in the preceding 12 months.
3. Current unstable or inadequately treated medical illness with the exception of current depression.
4. Recently started taking a CANMAT-recommended treatment for the management of acute bipolar depressive episode, but has not had a trial for a minimum of 6 weeks with adequate doses.
5. Recently (i.e. within the past 8 weeks) began structured psychotherapy (i.e. cognitive-behavioral therapy, interpersonal psychotherapy, family-focused therapy, or interpersonal and social rhythm therapy).
6. Recently (i.e. within the past 8 weeks) started taking a stimulant medication. Concomitant treatment with stimulant medication is acceptable provided that the dose has been stable for a minimum of 8 weeks and is taken as prescribed by a physician.
7. Current use of clozapine, tricyclic antidepressants, monoamine oxidase inhibitors, and first-generation antipsychotics.
8. A history of non-response or intolerance to CBD.
9. Current or past month daily use of CBD, or any product or drug that contains CBD. Occasional users will be included if they agree to refrain from using during the trial.
10. A history of non-response to electroconvulsive therapy for the current depressive episode.
11. A current diagnosis of other primary psychiatric disorders as assessed by a study investigator to be primary and causing greater impairment than BD.
12. A lifetime history of a primary psychotic disorder (e.g. schizoaffective disorder, bipolar subtype) according to DSM-5 criteria.
13. Patients who have met the DSM-5 criteria for a substance use disorder (except for nicotine or caffeine) within the past 6 months.
14. Significant active suicidal ideation (as evidenced by MADRS suicide item ≥ 4).
15. Pregnancy or lactation.
16. Liver function tests (AST and ALT) three times the upper limit of normal.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in depressive symptoms in bipolar patients treated with Cannabidiol vs Placebo adjunctive therapy | 6 weeks
  The Montgomery Asberg Depression Rating Scale (MADRS) will be used to measure change in depressive symptoms from baseline to endpoint. Scores range from 0 to 60, and lower scores reflect better clinical outcomes.

SECONDARY OUTCOMES:
Response rates | 6 weeks
  Response rates are defined as patients showing ≥50% reduction in MADRS scores.
Remission rates | 6 weeks
  Remission rates are defined as MADRS ≤ 10 and YMRS ≤ 8 at endpoint.
Treatment-emergent manic/hypomanic events | 6 weeks
  The Young Mania Rating Scale (YMRS) will be used to determine the presence of any treatment-emergent manic or hypomanic events from baseline to endpoint. Scores range from 0 to 60, and lower scores reflect better clinical outcomes.
Objective depressive symptoms | 6 weeks
  The 21-item Hamilton Depression Rating Scale (HAM-D 21) will be used to measure change in objective depressive symptoms from baseline to endpoint. Scores range from 0 to 62, and lower scores reflect better clinical outcomes.
Subjective depressive symptoms | 6 weeks
  The Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) and the Dimensional Anhedonia Rating Scale (DARS) will be used to measure change in subjective depressive symptoms from baseline to endpoint. Lower scores on the QIDS-SR reflect better clinical outcomes; higher scores on the DARS reflect better clinical outcomes.
Objective anxiety symptoms | 6 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) will be used to measure change in objective anxiety symptoms from baseline to endpoint. Scores range from 0 to 56 and lower scores reflect better clinical outcomes.
Subjective anxiety symptoms assessed by STAI | 6 weeks
  The State-Trait Anxiety Inventory (STAI) will be used to measure change in subjective anxiety symptoms. Lower scores on the STAI reflect better clinical outcomes.
Subjective anxiety symptoms assessed by GAD-7 | 6 weeks
  The Generalized Anxiety Disorder 7-item (GAD-7) will be used to measure change in subjective anxiety symptoms. Lower scores on the GAD-7 reflect better clinical outcomes.
Overall psychiatric status | 6 weeks
  The Clinical Global Impression - severity & change scales will be used to measure change in global severity and global improvement in symptoms from baseline to endpoint. Scores range from 3 to 42, and higher scores reflect worsening in overall psychiatric status.
Psychotic symptoms | 6 weeks
  The Positive and Negative Syndrome Scale (PANSS) will be used to measure change in psychotic symptoms from baseline to endpoint. Scores range from 7 to 49, and lower scores reflect better clinical outcomes.
Subjective cognitive functioning | 6 weeks
  The Cognitive Complaints in Bipolar Disorder Risk Assessment (COBRA) and the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function scale will be used to measure change in subjective cognitive functioning from baseline to endpoint. COBRA scores range from 0 to 48, and lower scores reflect better outcomes; PROMIS cognitive function scale scores range from 8 to 40, and higher scores reflect better outcomes.
Objective cognitive functioning | Week 6
  The Screen for Cognitive Impairment in Psychiatry (SCIP) will be used to measure change in objective cognitive functioning from baseline to endpoint. Higher scores reflect better outcomes.
Sleep quality | 6 weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used to measure changes in sleep quality and disturbance from baseline to endpoint. Lower scores reflect better sleep quality.
Suicidal thoughts and behaviours | 6 weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to measure change in suicidal thoughts and behaviours from baseline to endpoint. Scores range from 0 to 37, and lower scores reflect better clinical outcomes.
Quality of Life assessed by QoL.BD | 6 weeks
  The Brief Quality of Life in Bipolar Disorder (QoL.BD) will be used to measure change in quality of life from baseline to endpoint. Higher scores reflect higher quality of life.
Daily functioning | 6 weeks
  The Functioning Assessment Short Test (FAST) will be used to measure change in daily functioning from baseline to endpoint. Lower scores reflect better daily functioning.
Health services utilization | 6 weeks
  A healthcare utilization diary will be used to measure improvement in health services utilization from baseline to endpoint.
Adverse events | 6 weeks
  Adverse events will be measured objectively using an open-ended form and subjectively using the Frequency, Intensity, and Burden of Side Effects Rating (FIBSER). FIBSER scores range from 0 to 18, and lower scores reflect better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi N Yatham, MBBS, MRCPsy, Principal Investigator — University of British Columbia, Department of Psychiatry
Locations (6):
- Canada (6):
  - UBC Mood Disorders Centre, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Providence Care Hospital, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - Douglas Mental Health University Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No